CLINICAL TRIAL: NCT04748757
Title: Annexin A5 in Patients With Severe COVID-19 Disease: A Single Centre, Randomized, Double-blind, Placebo-controlled Pilot Trial
Brief Title: Annexin A5 in Patients With Severe COVID-19 Disease
Acronym: AX-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Ministry of Colleges and Universities (Unknown); London Health Sciences Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REDA-10122
Record Dates: First submitted 2021-02-02; First posted 2021-02-10 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Coronavirus Infection; Sepsis
MeSH Terms: conditions — Coronavirus Infections; Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Normal saline, 50 ml infusion over 30 minutes every 12 hours for 7 days
  Interventions: Drug: Placebo
- Low dose (Experimental): 50 microg/kg SY-005 in 50 ml saline infused over 30 minutes every 12 hours for 7 days
  Interventions: Drug: recombinant human annexin A5
- High dose (Experimental): 100 microg/kg SY-005 in 50 ml saline infused over 30 minutes every 12 hours for 7 days
  Interventions: Drug: recombinant human annexin A5

INTERVENTIONS:
Drug: recombinant human annexin A5 — recombinant human annexin A5, manufactured as SY-005
  Other Names: SY-005
  Arms: High dose; Low dose
Drug: Placebo — Normal saline 50 ml
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled trial comparing 2 doses of SY-005 (recombinant human Annexin A5) to placebo in patients with severe coronavirus 2019 disease in a single hospital centre with 2 intensive care units

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years
2. Positive test for SARS-CoV-2 virus (anytime during current illness episode)
3. Admitted to intensive care for organ failure support (at least one of vasopressor, non-invasive or invasive ventilation)

Exclusion Criteria:

1. Known allergy to any of the ingredients or components of the investigational product
2. Known pregnancy
3. Moribund and not expected to survive beyond 24 hours
4. Known or suspected risk for serious bleeding complications (note that Disseminated Intravascular Coagulopathy (DIC) is an expected finding in patient with sepsis and COVID-19 disease and is not an exclusion criterion on its own)
5. Acute or chronic renal failure (dialysis dependent)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-04-03 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Enrollment | 12 months
  Participants enrolled per site per month with success defined as enrollment >= 50% of screened eligible patients
Protocol adherence | 7 days
  Delivery of investigational product within 1 hour of scheduled dose; success defined as >= 90%
Data completeness | 12 months
  Case Report Forms completed with <10% missing data after verification and monitoring

SECONDARY OUTCOMES:
Organ failure | 30 days
  Sequential Organ Failure Assessment (SOFA) at 30 days; range 0 (normal) to 24
Organ function at end of treatment measured with SOFA | 7 days
  SOFA at end of treatment (EOT)
Organ function at end of treatment measured with Multiple Organ Dysfunction Score (MODS) | 7 days
  MODS at end of treatment (EOT); range 0 (normal) to 24
Individual organ function scores at EOT measured with SOFA | 30 days
  SOFA for individual organ systems
Individual organ function scores at 30 days measured with SOFA | 30 days
  SOFA for individual organ systems
Individual organ function scores at EOT measured with MODS | 30 days
  MODS for individual organ systems
Individual organ function scores at 30 days measured with MODS | 30 days
  MODS for individual organ systems
Plasma annexin A5 levels daily days 1-8 (treatment period) and on day 14 | 14 days
  Annexin A5 will be measured daily during treatment and on day 14
Mortality at 60 days | 60 days
  All cause mortality
Hospital mortality | 60 days
  Hospital mortality censored at 60 days
Ventilator-free days | 30 days
  Days alive and off ventilator at 30 days
ICU-free days | 30 days
  Days alive and not in ICU at 30 days
Number of participants with persistent organ dysfunction | 30 days
  MODS score greater or equal to 2 in any organ system at day 30
Number of serious adverse events (SAE) | 60 days
  SAE
Maximum plasma concentration (Cmax) of annexin A5 (SY-005) | 1 day
  Pharmacokinetic profile on day 1
Elimination half-life of annexin A5 (SY-005) | 1 day
  Pharmacokinetic profile on day 1
Number of participants with anti-annexin A5 antibodies | 21 days
  Anti-annexin A5 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Martin, MD, MSc, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Information and data sharing will be considered on individual basis at conclusion of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: To be evaluated on individual basis

REFERENCES:
- [Derived] Tschirhart BJ, Lu X, Mokale Kognou AL, Martin CM, Slessarev M, Fraser DD, Leligdowicz A, Urquhart B, Feng Q. Pharmacokinetics of recombinant human annexin A5 (SY-005) in patients with severe COVID-19. Front Pharmacol. 2024 Jan 10;14:1299613. doi: 10.3389/fphar.2023.1299613. eCollection 2023. PMID 38269269